CLINICAL TRIAL: NCT06958900
Title: Effect of Malignancy on Morbidity and Mortality in Left-sided Emergency Colorectal Resections
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasir Musa Kesgin, MD, General Surgery Specialist, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2024-166
Record Dates: First submitted 2025-01-24; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-01

CONDITIONS: Emergency Abdominal Surgery; Colorectal Surgery; Acute Diverticulitis; Volvulus
Keywords: Colorectal Cancer; Emergency Surgery; Morbidity; Mortality
MeSH Terms: conditions — Intestinal Volvulus; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Emergency Left-Sided Colorectal Resections: Patients in a single center underwent emergency left-sided colorectal resection due to benign or malign colorectal pathology

SUMMARY:
Patients who underwent emergency left sided colorectal resection in a single center between January 2023 and May 2024 were included. Demographics, Charlson comorbidity index, perforation, duration of surgery, primary anastomosis or end colostomy preference and benign or malign etiologies were examined. Morbidity was defined as Clavien Dindo grade III or higher complication. Risk factors for both morbidity and mortality were first evaluated with univariate analyzes. Then multivariable logistic regression tests were performed for both morbidity and mortality.

DETAILED DESCRIPTION:
Patients in a single center between January 2023 and May 2024 were included in this retrospective observational study. Included patients who were 18 years old or older and underwent emergency left-sided colorectal resection due to isolated colorectal pathology. Patients with diseases originated from a colonic segment proximal to left colon, surgeries performed for combined organ pathologies for various benign and malignant causes and those undergoing reoperation caused by complication of elective abdominal surgery were excluded Data of patients obtained via the hospital software system. Demographic data, Charlson comorbidity index (CCI) score and baseline characteristics, operative and postoperative results, primary anastomosis or end colostomy preference, length of hospital stay, presence of perforation and and benign or malign etiologies were investigated. Morbidity was defined as Clavien Dindo grade III or higher complication.

Risk factors for both morbidity and mortality were first evaluated using univariate analyzes. In univariate analysis for morbidity, patients divided two subgroups as patient with morbidity and the others without morbidity. After that these two subgroups compared in terms of all variables. For univariate mortality analysis also, patients divided again according to dying in first 90 days postoperatively or not. After that these mortality and alive subgroups analysed in terms of all variables. Pearson Chi Square, Student's t-test and Mann Whitney U tests were used when appropriate. Decision for normal distribution was given according to Kolmogorov- Smirnov test. Values for normally distributed variables expressed as mean±standard deviation (SD). Categorical variables are expressed as number and percentage. The variables that not showed a normal distribution expressed as median and 25-75 interquartile range values. The effects of risk factors on morbidity and mortality were expressed as the odds ratio with their 95% confidence intervals (CI). Statistical significance level was set at 0.05. The data were compiled and analyzed using the software SPSS for Windows, version 29.0 (SPSS, Chicago, IL)

ELIGIBILITY:
Inclusion Criteria:

* Patients who were 18 years old or older and underwent emergency left-sided colorectal resection due to isolated colorectal pathology

Exclusion Criteria:

* Patients with diseases originated from a colonic segment proximal to left colon, surgeries performed for combined organ pathologies for various benign and malignant causes and those undergoing reoperation caused by complication of elective abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were 18 years old or older and underwent emergency left-sided colorectal resection due to isolated colorectal pathology
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Morbidity | Postoperative 30 days
  Morbidity was defined as Clavien Dindo grade III or higher postoperative complication.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)